CLINICAL TRIAL: NCT03903939
Title: Efficacy and Safety of 72-hour Infusion of Prostacyclin (1 Nanogram(ng)/Kilogram(kg)/Minute(Min)) in Trauma Patients With Haemorrhagic Shock Induced Endotheliopathy.
Brief Title: Infusion of Prostacyclin vs Placebo for 72-hours in Trauma Patients With Haemorrhagic Shock Suffering From Organ Failure
Acronym: SHINE-TRAUMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pär Johansson (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Pär Johansson, Clinical professor, Head of Section for Transfusion Medicine, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHINE-TRAUMA; 2019-000936-24 (EudraCT Number)
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multi Organ Failure
Keywords: Trauma patients; Shock-induced endotheliopathy
MeSH Terms: conditions — Multiple Organ Failure | interventions — Iloprost; Methods; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both patient, investigator and outcome assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iloprost (Experimental): Patients randomized to active treatment (n = 110 patients) will receive continuous infusion of iloprost for 72 hours after inclusion or until discharge to ward or death, whichever comes first
  Interventions: Drug: Iloprost
- Placebo (Placebo Comparator): Patients randomized to placebo treatment (n= 110 patients) will receive continuous infusion of isotonic saline (equal volume) for 72 hours after inclusion or until discharge to ward or death, whichever comes first.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Iloprost — continuously infusion for 72 hours 1 ng/kg/min
  Other Names: Intervention
  Arms: Iloprost
Drug: Isotonic saline — continuously infusion for 72 hours equal volume to Iloprost
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A multicenter, randomized (1:1, iloprost: placebo), placebo controlled, blinded, investigator-initiated phase 2b trial in trauma patients with haemorrhagic shock and shock induced endotheliopathy (SHINE), investigating the efficacy and safety of continuous intravenous administrating of iloprost (1 ng/kg/min) versus placebo for 72-hours, in a total of 220 patients.

The study hypothesis is that iloprost may be beneficial as an endothelial rescue treatment as it is anticipated to deactivate the endothelium and restore vascular integrity in trauma patients with haemorrhagic shock (SHINE) suffering from organ failure caused by endothelial breakdown, ultimately improving survival.

DETAILED DESCRIPTION:
The main objective in this trial is to investigate whether continuous infusion of iloprost at a dose of 1 ng/kg/min for 72-hours is safe and significantly increase the number of intensive care unit (ICU) free days, within 28 days from admission compared to infusion of placebo in trauma patients with haemorrhagic shock and SHINE.

Patients are presented at the investigator site in an acute critical condition and therefore informed consent will be obtained from a scientific guardian. Next-of-kin and subsequently the patient will co-sign as soon as possible. During the trial additional blood samples will be obtained daily for the first 72 hours. Patients will be observed and assessed continuously. During the extended follow up period at day 28 and 90, no contact will be made to the patient, but the data will be collected from department/hospital databases to establish length of stay and potential mortality.

The trial is conducted in accordance with the Helsinki 2 declaration and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use, Guideline for Good Clinical Practice (ICH-GCP) and in compliance with the protocol. As part of the quality assurance site monitoring will be performed by an independent GCP-Unit including source data verification. Standard Operation Procedure to address protocol specific procedures such as data collection and adverse event reporting are developed.

The power calculation is based on not yet published data from the following trial 'Implementing Treatment Algorithms for the Correction of Trauma Induced Coagulopathy (iTACTIC)' [NTC 02593877] having the same in- and exclusion criteria as the present trial. The number of ICU free days within 30-days from admission is chosen as the primary endpoint and a clinically relevant increase in ICU free days within 28-days of 30% with α 0.05, power 0.85 will require 107 patients in each 1:1 randomization group. We plan on including 110 patients in each group and 220 in total. The final statistical analysis plan will be published before the last patient is included in the trial and analysis of the data from the randomized trial will be performed by Theis Lange, Associate Professor, Section of Biostatistics, Department of Public Health, University of Copenhagen.

The primary end point will be analyzed using linear regression adjusted for site. Effect size will be summarized using adjusted mean differences with confidence intervals based on robust standard errors as residuals are not expected to be normally distributed. The same analysis will be employed to continuous secondary outcomes. All-cause mortality will be further illustrated using Kaplan-Meier curves. All analysis will be conducted following the intention to treat principle (this will be the primary analysis) and per-protocol. In addition, the following patient subgroup will also be analyzed separately:

• Patients with traumatic brain injury

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Present with clinical signs of hemorrhagic shock (defined by systolic blood pressure <90 millimetre of mercury (mmHg) or use of pre-hospital blood transfusion).
* Activation of local massive transfusion protocol and initiation of the first transfusion after admission.
* Randomised within 5 hours of injury and 3 hours of admission to the emergency department of the participating trial site.
* Consent is provided on behalf of incapacitated patients by Scientific Guardian

Exclusion Criteria:

* Withdrawal from active therapy
* Known hypersensitivity to Iloprost.
* Pregnancy (non-pregnancy confirmed by patient having a negative urine or plasma choriogonadotropin (hCG) or being postmenopausal defined as females at 60 years old and beyond)
* Known severe heart failure (New York Heart Association (NYHA) class IV)
* Suspected acute coronary syndrome
* Estimated weight < 40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
ICU free days | 28 days after admission
  Defined as the number of days spend alive out of the ICU to day 28. Patients who dies on or prior to day 28 during their initial ICU stay are assigned zero in ICU free days

SECONDARY OUTCOMES:
All-cause mortality | 90 days after admission
  Vital status of the patient at day 28 and 90.
Hospital length of stay | 90 days after admission
  Defined as the total number of days admitted to the hospital until day 90
Vasopressor free days | 28 days after admission
  The number of calendar days between admission and 28 days later that the patients is alive and without the use of vasopressor therapy
Ventilator free days | 28 days after admission
  The number of calendar days between admission and 28 days later that the patients is alive and without the use of mechanical ventilation. Ventilator meaning mechanical ventilation via endotracheal or tracheostomy tube, except those intubated solely for a procedure. Non-invasive mechanical ventilation will not be included.
Renal replacement free days | 28 days after admission
  The number of calendar days between admission and 28 days later that the patient is alive and without renal replacement therapy. Patients with chronic renal replacement therapy initiated prior to the current admission will not be included unless worsen.
Serious adverse reactions | 4 days after randomization
  Number of serious adverse reactions (SARs) in the 2 arms. SARs is defined as any untoward medical reactions that at any dose results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalization, results in persistent or significant disability or incapacity or is a congenital anomaly or birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Pär I Johansson, MD, MPA, Study Director — University of Copenhagen (Rigshospitalet)
Locations (5):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet (University of Copenhagen), Copenhagen
  - Odense University Hospital, Odense
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansson PI, Eriksen CF, Schmal H, Gaarder C, Pall M, Henriksen HH, Bovbjerg P, Lange T, Naess PA, Nielsen C, Kirkegaard H, Stensballe J. Efficacy and safety of iloprost in trauma patients with haemorrhagic shock-induced endotheliopathy-Protocol for the multicentre randomized, placebo-controlled, blinded, investigator-initiated shine-trauma trial. Acta Anaesthesiol Scand. 2021 Apr;65(4):551-557. doi: 10.1111/aas.13776. Epub 2021 Jan 11. PMID 33393084
- See also: Publication of results — https://pubmed.ncbi.nlm.nih.gov/37962189/